CLINICAL TRIAL: NCT02967276
Title: Phase II Trial, Open Label, Clinical Activity of Metformin in Combination With High-dose of Dexamethasone (HDdexa) in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Clinical Activity of Metformin With High-dose of Dexamethasone in Relapse Multiple Myeloma
Acronym: METDEXA-MM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Ademar Dantas da Cunha Júnior, Principal investigator, University of Campinas, Brazil
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: METDEXA-MM
Record Dates: First submitted 2016-11-04; First posted 2016-11-18 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2016-11

CONDITIONS: Multiple Myeloma
Keywords: Metformin; Dexamethasone; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin and HDdexamethasone (Experimental): Metformin XR is initially administered at a dose of 500mg / daily by oral administration for 7 days. Patients who have a good tolerance (lack of adverse events of grade 3 or 4) may be staggered metformin dose to 2500 mg / day.
  Patients in turn receiving dexamethasone pulse prescription (HDdex). A dose of dexamethasona 40 mg / day taken in a daily for four days every 8 days from 1st to 2nd cycle every 35 days and 1x per week for 4 weeks every 28 days from the 3rd to 6th cycle. The dose will be administered at 4 mg tablets, which are to be swallowed whole by 30 minutes after a meal. Patients over age 75 used 20 mg / day.
  Interventions: Drug: Metformin XR; Drug: Dexamethasone

INTERVENTIONS:
Drug: Metformin XR — 500 mg tablet: They take 1-5 tablets of 500 mg after dinner. Starting dose of Metformin XR 500 mg. It will have an increase of 500 mg/day each week up to the maximum tolerance from the 2500 mg / day, during the 6 cycles.
  Other Names: Glifage XR
Drug: Dexamethasone — 4 mg tablet: Patients will use 40 mg per day. They take 5-10 tablets 4mg after breakfast and lunch. Patients over age 75 will use 20 mg / day.
  Other Names: Decadron

SUMMARY:
This phase II trial study assessing the activity of metformin when given together with high dose of dexamethasone in treating patients with multiple myeloma (MM) that has relapse or refractory to previous treatment. High dose of dexamethasone (HDdexa) is used to treat relapse/refractary patients with myeloma and metformin also demonstrated synergistic activity with dexamethasone to eradicate MM cells in vitro and in vivo. Metformin hydrochloride, used for diabetes, may also help kill tumor cells. Giving dexamethasone with metformin may kill more MM cells and increase the response rate to HDdexa.

DETAILED DESCRIPTION:
Phase II trial, open label, clinical activity of metformin combination with high-dose dexamethasone (HDdexa) in patients with multiple myeloma relapsed-refractory.

If you are found to be eligible to take part in this study, metformin will be given continuously until completion of the treatment, disease progression, severe toxicity or intolerance. The same duration of treatment will be applied to dexamethasone.

The treatment will be initiated with dexamethasone (40 mg daily for 4 days on D1-D4, D9-D12 and D17-D20) Before starting the HDDexa investigators will obtain blood and bone marrow samples for evaluation of response to the disease using biomarkers of multiple myeloma. On day 1, the patients will begin metformin XR (500mg daily with the evening meal) with gradual increase in the dose - 500 mg per week up to a maximum of 2.5 g / day if no toxicity grade ≥ 2 . Each cycle will be reset every 35 days in the 1st and 2nd cycle and every 28 days from 3rd to 6th cycle. Patients who maintained clinical response to treatment after the first cycle should use the drugs for 6 cycles, or until progression or unacceptable toxicity. Oral dexamethasone (40 mg) is administered on days 1 to 4, 9 to 12 and 17 to 20 the first and second (cycles of 35 days) and on days 1, 8, 15 and 22 of the third to sixth (cycle 28d), for a period of 190 days of treatment. Patients over 75 years will use 20 mg / day instead of 40 mg / day.

Patients will be submitted to collection of tissues: blood and bone marrow to evaluate the response to disease through multiple myeloma biomarkers before the first cycle, 4th and 5th cycle of treatment to assess the response according to IMWG criteria: blood count, creatinine , calcium, lactate dehydrogenase (LDH); Beta2 microglobulin; C-reactive protein (CRP) and erythrocyte sedimentation rate (ESR); Immunoelectrophoresis and immunofixation of the proteins in serum and urine 24 hours; 24h proteinuria; Myelogram and bone marrow biopsy (BMO) and Immunophenotyping. Clinical and laboratory exams will be conducted at the beginning and every 35 days on first 2 cycles every 28 days until the 6th cycle.

Safety assessments will include history and physical examination, electrocardiography, blood count, biochemical tests (including glucose and glycated Hb) and pulse oximetry.

Toxic effects will be analyzed according to the National Cancer Institute Common Toxicity Criteria for Adverse Events, version 4 (NCI CTCAE v4).

This is an investigational study. Dexamethasone is FDA approved and commercially available for the treatment of many inflammatory diseases. Metformin is FDA approved and commercially available for the treatment of diabetes mellitus. The combination of these drugs to treat multiple myeloma is investigational.

Up to 28 patients will take part in this study. This is a multicenter study, and will take place in the clinical research center at the Clinical Hematology of the Clinical Hospital, University of Campinas-UNICAMP and at the Cascavel Cancer Hospital - UOPECCAN. This study will be coordinated by the Hemocentro-UNICAMP

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years;
* Multiple myeloma patients relapsed or refractory to two lines prior to treatment [at least one line using bortezomib or prior treatment with a suitable alkylating agent (at least six cycles of treatment with alkylating or progressive disease after at least two cycles of treatment with alkylating or treatment with alkylating received as part of a stem cell transplant)];
* Patients should have failed (progressive disease at or before 60 days of treatment, disease progression ≤6 months after achieving partial response or intolerance to bortezomib) to treatment with bortezomib;
* Patients with oral access to medicines;
* ECOG ≤ 2;
* Blood count: hemoglobin ≥8 g / dL; absolute neutrophil count ≥500 / mm3 and platelet count ≥30.000 / mm3, glomerular filtration rate (GFR) ≥60ml / min and adequate liver function (AST or ALT at levels 3x upper limit of normal, bilirubin in levels no greater than 2x the upper limit of normal, negative pregnancy test before study initiation or accept contraceptive use.

Exclusion Criteria:

* Patients with known hypersensitivity and / or prior therapy with metformin or its excipients;
* Diabetes mellitus who require insulin use and other oral hypoglycemic agents; patients with a history of hyperglycemia induced by steroids can be entered since HbA1C in screening visit is <8%;
* leptomeningeal or brain metastases symptomatic or untreated, or spinal cord compression;
* Known human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) (with the exception treated or cured chronic HBV and HCV infection, who will be allowed);
* Patients who are using another study medication or who have received drug under study for less than 4 weeks;
* It is allowed concomitant treatment with bisphosphonates; however, treatment should be started before the first dose of study therapy;
* it is not allowed to use of all herbal supplements during the study (including, but not limited to, St. John's wort, kava, None, gingko biloba, dehydroepiandrosterone [DHEA], or ginseng). megestrol acetate (Megace) or medroxyprogesterone if used as an appetite stimulant is permitted;
* Uncontrolled situations by intercurrent disease, including, but not limited to, infection ongoing and active, refractory systemic hypertension, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric / social disease that would limit compliance with the requirements of study;
* Previous Neoplasms, except skin cancer for over two years;
* Patients who are pregnant or breastfeeding.
* Any major surgery, extensive radiation therapy, chemotherapy delayed toxicity, biological therapy, chemotherapy or immunotherapy within 28 days before study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Response Rate (RR) | From the date of randomization to the date of the first major documented response (CR, PR or MR) that occurs, evaluated up to 35 days after the completion of 6th treatment cycles or if the response occurs earlier.
  the RR to metformin and HDdexa schedule including: complete (CR), partial (PR) and minimal (MR) response in patients with relapsed/refractory multiple myeloma criteria for defining response according to the International Myeloma Working Group (IMWG): CR: Negative immunofixation of serum and urine, and Disappearance of any soft tissue plasmacytomas, and below of 5% Plasma Cells in bone marrow. PR: above or equal 50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by 90% or 200 mg/24 hours. MR: above or equal 25% but below or equal 49% reduction of serum M-protein and reduction in 24-hour urine M-protein by 50%-89%.

SECONDARY OUTCOMES:
Time to progression (TTP) during treatment with metformin and HDdexa according to criteria for defining response of the International Myeloma Working Group (IMWG) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  TTP:Duration from start of treatment to disease progression, with deaths from causes other than progression censored.
Duration of response (DOR) during treatment with metformin and HDdexa according to criteria for defining response of the International Myeloma Working Group (IMWG) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  DOR: Duration from first observation of partial response (PR) to the time of disease progression, with deaths from causes other than progression censored.
Event free survival (EFS) during treatment with metformin and HDdexa according to criteria for defining response of the International Myeloma Working Group (IMWG) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  EFS: Duration from start of the treatment to disease progression or death (regardless of cause of death), whichever comes first. The definition of EFS used is the same as PFS.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - UOPECCAN - Hospital do Câncer de Cascavel, Cascavel, Paraná
  - Hemocentro - Hospital de Clínicas - State University of Campinas (UNICAMP), Campinas, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zi FM, He JS, Li Y, Wu C, Yang L, Yang Y, Wang LJ, He DH, Zhao Y, Wu WJ, Zheng GF, Han XY, Huang H, Yi Q, Cai Z. Metformin displays anti-myeloma activity and synergistic effect with dexamethasone in in vitro and in vivo xenograft models. Cancer Lett. 2015 Jan 28;356(2 Pt B):443-53. doi: 10.1016/j.canlet.2014.09.050. Epub 2014 Oct 8. PMID 25305450
- [Background] Jagannathan S, Abdel-Malek MA, Malek E, Vad N, Latif T, Anderson KC, Driscoll JJ. Pharmacologic screens reveal metformin that suppresses GRP78-dependent autophagy to enhance the anti-myeloma effect of bortezomib. Leukemia. 2015 Nov;29(11):2184-91. doi: 10.1038/leu.2015.157. Epub 2015 Jun 25. PMID 26108695
- [Background] Wu W, Merriman K, Nabaah A, Seval N, Seval D, Lin H, Wang M, Qazilbash MH, Baladandayuthapani V, Berry D, Orlowski RZ, Lee MH, Yeung SC. The association of diabetes and anti-diabetic medications with clinical outcomes in multiple myeloma. Br J Cancer. 2014 Jul 29;111(3):628-36. doi: 10.1038/bjc.2014.307. Epub 2014 Jun 12. PMID 24921909
- [Background] Dowling RJ, Niraula S, Stambolic V, Goodwin PJ. Metformin in cancer: translational challenges. J Mol Endocrinol. 2012 Mar 29;48(3):R31-43. doi: 10.1530/JME-12-0007. Print 2012 Jun. PMID 22355097